CLINICAL TRIAL: NCT07342946
Title: Effects of a Mediterranean Diet and Synbiotic Supplementation on Anthropometric and Biochemical Parameters and Quality of Life in Obese Women With Polycystic Ovary Syndrome
Brief Title: The Effects of the Mediterranean Diet and Synbiotics in Polycystic Ovary Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Aysenur Emirhuseyinoglu Calik, Research Assistant, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-22686390-050.99-78501
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: synbiotics; pcos; diet; nutrition
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in this arm will receive a hypocaloric Mediterranean diet in addition to a placebo for a period of 8 weeks.
  Interventions: Other: Placebo
- Synbiotics (Active Comparator): Participants in this arm will receive a hypocaloric Mediterranean diet in addition to synbiotic supplementation for a period of 8 weeks.
  Interventions: Dietary Supplement: Synbiotic Supplement

INTERVENTIONS:
Dietary Supplement: Synbiotic Supplement — Participants in this arm will receive a hypocaloric Mediterranean diet in addition to synbiotic supplementation for a period of 8 weeks.
  Other Names: Mediterrenean Diet
  Arms: Synbiotics
Other: Placebo — Participants in this arm will receive a hypocaloric Mediterranean diet in addition to a placebo for a period of 8 weeks.
  Other Names: Mediterrenean Diet
  Arms: Placebo

SUMMARY:
This study will look at whether a reduced-calorie Mediterranean-style eating plan, together with a synbiotic supplement, can improve health measures and quality of life in women who have polycystic ovary syndrome (PCOS) and are overweight or have obesity. Participants will be assigned by chance (like flipping a coin) to receive either the synbiotic supplement or a placebo (a look-alike product with no active ingredients). All participants will follow the same reduced-calorie Mediterranean diet for 8 weeks. The study team will measure body composition and weight-related measurements, and will collect blood samples to evaluate selected laboratory markers before and after the 8-week period. Participants will also complete the PCOSQ-50 quality-of-life questionnaire before and after the intervention. The goal is to better understand the possible role of synbiotic supplementation alongside dietary treatment in PCOS.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, single-blind clinical trial is designed to evaluate the effects of a hypocaloric Mediterranean diet combined with synbiotic supplementation on anthropometric measurements, biochemical parameters, and quality of life in overweight and obese women diagnosed with polycystic ovary syndrome (PCOS). Eligible participants will be randomly assigned to one of two study arms: a synbiotic supplementation group or a placebo group. Both groups will follow the same hypocaloric Mediterranean diet throughout the 8-week intervention period.

Anthropometric assessments, including body weight, body mass index, waist circumference, and body composition, will be performed at baseline and at the end of the intervention. Biochemical parameters will be evaluated through blood samples collected at baseline and after 8 weeks. Quality of life will be assessed using the PCOSQ-50 Quality of Life Questionnaire at both time points.

The study aims to determine whether the addition of synbiotic supplementation to a hypocaloric Mediterranean diet provides additional benefits in the management of PCOS-related metabolic parameters and quality of life compared with dietary intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women who are overweight or obese, with a body mass index (BMI) between 25 and 35 kg/m²
* Aged 18 to 45 years (reproductive age)
* Diagnosed with polycystic ovary syndrome (PCOS)

No underlying metabolic diseases, including type 2 diabetes mellitus, hypertension, diagnosed anemia, or any other metabolic condition requiring a special diet

Exclusion Criteria:

* Pregnancy or breastfeeding within the past 6 months
* Presence of comorbid conditions, including kidney, liver, or cardiovascular disease, gout, hyperuricemia, or other related disorders
* Use of oral contraceptives
* Following a special dietary treatment or a hypocaloric diet within the last 3 months
* Occasional or current use of medications that may affect fluid balance, including diuretics and laxatives
* Participants will be withdrawn from the study in case of abnormal biochemical parameters, non-adherence to the prescribed diet, or failure to comply with the supplementation protoco

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 32 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | From enrollment to the end of treatment at 8 weeks
  Changes in body weight measured in kilograms using the Tanita MC-780 bioelectrical impedance analysis (BIA) device at baseline and after the 8-week intervention.
Change in body mass index (BMI) | From enrollment to the end of treatment at 8 weeks
  Changes in body mass index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m²), with body weight measured using the Tanita MC-780 bioelectrical impedance analysis (BIA) device at baseline and after the 8-week intervention.
Change in body composition | From enrollment to the end of treatment at 8 weeks
  Changes in body composition parameters, including fat mass and fat-free mass, assessed using the Tanita MC-780 bioelectrical impedance analysis (BIA) device at baseline and after the 8-week intervention.
Change in waist circumference | From enrollment to the end of treatment at 8 weeks
  Changes in waist circumference measured in centimeters using a non-elastic measuring tape at baseline and after the 8-week intervention.
Change in hip circumference | From enrollment to the end of treatment at 8 weeks
  Changes in hip circumference measured in centimeters using a non-elastic measuring tape at baseline and after the 8-week intervention.

SECONDARY OUTCOMES:
Change in insulin resistance (HOMA-IR) | From enrollment to the end of treatment at 8 weeks
  Changes in insulin resistance assessed using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting plasma glucose and fasting insulin levels. A HOMA-IR value below 2.5 will be considered indicative of the absence of insulin resistance. Measurements will be performed at baseline and after the 8-week intervention.
Change in fasting blood glucose | From enrollment to the end of treatment at 8 weeks
  Changes in fasting blood glucose levels measured in mg/dL from venous blood samples collected at baseline and after the 8-week intervention.
Change in lipid profile | From enrollment to the end of treatment at 8 weeks
  Changes in serum lipid profile parameters, including high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), triglycerides (TG), and total cholesterol, measured in mg/dL from venous blood samples collected at baseline and after the 8-week intervention.
Change in follicle-stimulating hormone (FSH) levels | From enrollment to the end of treatment at 8 weeks
  Changes in serum follicle-stimulating hormone (FSH) levels measured from venous blood samples collected at baseline and after the 8-week intervention.
Change in luteinizing hormone (LH) levels | From enrollment to the end of treatment at 8 weeks
  Changes in serum luteinizing hormone (LH) levels measured from venous blood samples collected at baseline and after the 8-week intervention.
Change in quality of life | From enrollment to the end of treatment at 8 weeks
  Changes in quality of life assessed using the Polycystic Ovary Syndrome Quality of Life Questionnaire (PCOSQ-50), a validated disease-specific instrument consisting of 50 items across six domains: psychosocial and emotional well-being, fertility, sexual function, obesity and menstrual irregularity, hirsutism, and coping with the disease. Each item is scored on a 5-point Likert scale ranging from 1 (always) to 5 (never), resulting in a total score range of 50 to 250. Higher scores indicate better quality of life. Domain scores are calculated as the mean of the items answered within each domain, excluding unanswered items. Assessments will be performed at baseline and after the 8-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Sivri-Aydın, Study Director — Atlas University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hariri Z, Yari Z, Hoseini S, Abhari K, Sohrab G. Synbiotic as an ameliorating factor in the health-related quality of life in women with polycystic ovary syndrome. A randomized, triple-blind, placebo-controlled trial. BMC Womens Health. 2024 Jan 3;24(1):19. doi: 10.1186/s12905-023-02868-1. PMID 38172876
- [Background] Koyutürk, G., & Külünkoğlu, B. A. (2023). Polikistik Over Sendromu Yaşam Kalitesi-50 Ölçeği'nin Türkçe uyarlamasının geçerlik ve güvenirliği. Sağlık ve Yaşam Bilimleri Dergisi, 5(2), 63-70.